CLINICAL TRIAL: NCT02610946
Title: Do Technology Apps Improve Compliance in Adolescent Renal Transplant Recipients?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Ha Tran, Principle Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: StanfordU TeenTransplant
Record Dates: First submitted 2015-11-16; First posted 2015-11-20 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Kidney Transplantation
Keywords: pediatric; adolescent; compliance
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Paper-based (Placebo Comparator): Use of paper-based calenders, reminders, medication list, and blood pressure, fluid intake tracking methods in adolescent renal transplant care
  Interventions: Behavioral: Paper-based
- Electronic application (Experimental): Use of electronic apps (iphone or i-Pad mini) to determine whether it can improve compliance with transplant care and readiness to transition to adult care.
  Interventions: Behavioral: Electronic application

INTERVENTIONS:
Behavioral: Electronic application — Electronic application (app) based intervention to improve adolescent compliance with transplant care and readiness to transition to adult care.
  Arms: Electronic application
Behavioral: Paper-based — Paper-based intervention to improve adolescent compliance with transplant care and readiness to transition to adult care.
  Arms: Paper-based

SUMMARY:
The purpose of this study is to empower adolescent renal transplant recipients to fully understand their medical condition as well as to help them acquire the skills to maintain a healthy allograft well into adulthood. It is hoped that introducing technological applications (apps) will assist adolescents in managing medications, clinic appointments, lab appointments, and in tracking fluid intake, blood pressure, caloric intake, and exercise frequency. The investigators aim to improve adolescent post-renal transplant outcomes (increase medication adherence, lower clinic and laboratory no-show rate, lower blood pressure and BMI, maintain creatinine clearance, decrease proteinuria, decrease incidence of allograft rejection, decrease hospitalizations) as well as reduce cost.

DETAILED DESCRIPTION:
The research team as well and principal investigator will identify and verify patient eligibility. Patients who are unable to speak or converse via sign language will be excluded. All participants will need to provide informed written consent.

For recruitment and informed consent, the expected benefits, risks, and uncertainties will be discussed with participants and their families. Participants will be offered enrollment in either the randomized trial or a concurrent observational cohort, which may be more feasible for families who live further away and have alternative insurance plans (Kaiser). The results of the concurrent observational cohort can be reported at a later time.

Enrollment will begin in April 2015 and end in April 2016. This is to ensure that patients who may miss an appointment can still be recruited in the following months.

Baseline variables will be collected prior to randomization including questionnaire and baseline characteristics such as age, creatinine, weight, height, BMI, urine protein-to-creatinine ratio, donor specific antibody levels, and blood pressure will be recorded. Blood draws will be done per standard of care only and blood samples will not be stored for research purposes. Computer-generated random treatment assignments will be made based on permuted blocks (randomly generated blocks of 3).

The experimental arm will have all participants attend monthly renal transplant adolescent clinic where the participant will undergo a 25-question baseline questionnaire focusing on the participant's current knowledge of own medical condition, medications, medication dosage, insurance coverage, daily fluid goal, blood pressure goal, voiding schedule, etc.

During each clinic visit, the participant will take the questionnaire and review results with the transplant/research coordinator. The transplant/research coordinator will also assist the participant in updating medication list, medication schedule, lab schedule, clinic appointment schedule, pharmacy refill schedule etc. using an electronic device with downloadable mobile apps. The included apps will be MyFitnessPal, a calorie counter and exercise tracker, Blood Pressure Lite (Codulis) for blood pressure recording, and Med Coach (GreatCall, Inc), providing medication and appointment reminders. If the participant already has a personal i-Phone, the study coordinator will assist the participant add schedules to the calendar and help set alarms and reminders. The research coordinator will also help download free mobile apps that will log BP, fluid intake, caloric intake, and exercise duration. If the participant does not have an i-Phone, an i-Pad Mini will be provided and the transplant coordinator will assist with all that as stated above. The participant will be seen by a nephrologist, social worker, and psychologist.

The non-technological group participants will also attend monthly renal transplant adolescent clinic where he/she will undergo the same 25-question baseline questionnaire. During each clinic visit, the participant will take the questionnaire and review results with the research coordinator. The transplant coordinator will also assist the participant in updating medication list, medication schedule, lab schedule, clinic appointment schedule, pharmacy refill schedule etc. using paper calendar and pre-printed paper logs per the routine care protocol. The participant will also be seen by a nephrologist, social worker, and psychologist.

The primary measure is performance on monthly medical knowledge questionnaire, used as a surrogate marker for readiness to transition to adult care. Secondary measures include medication adherence measured by immunosuppression target drug levels, clinic and laboratory no-show rates, markers of graft function measured by blood pressure readings, BMI, creatinine clearance, urine protein-to-creatinine ratio, and episodes of rejections measured by donor specific antibodies, and pathologic findings of allograft biopsy. The study will end after the one year follow up period is completed. As the paper-based strategy is to function as a control, the investigators do not anticipate an early termination to the study, particularly since both groups provide more intervention than the current standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent patients between 12 and 18 years of age with kidney transplants seen at Lucile Packard Children's Hospital for their transplant care at least every 3 months.

Exclusion Criteria:

* Non-English speaking,
* significant cognitive delays,
* seen in clinic less often than every 3 months.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Compliance | 1 year
  Ability to adhere to medical recommendations of transplant care assessed by presence or absence of antibody-mediated rejection based on donor-specific antibody levels.

SECONDARY OUTCOMES:
Readiness to transition | 1 year
  Knowledge of transplant care and readiness to transition to adult care assessed by questionnaire of disease knowledge base taken at baseline and at end of study

CONTACTS AND LOCATIONS:
Overall Officials: Ha Tran, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University Hospital and Clinics, Palo Alto, California, United States

REFERENCES:
- [Derived] Mellon L, Doyle F, Hickey A, Ward KD, de Freitas DG, McCormick PA, O'Connell O, Conlon P. Interventions for increasing immunosuppressant medication adherence in solid organ transplant recipients. Cochrane Database Syst Rev. 2022 Sep 12;9(9):CD012854. doi: 10.1002/14651858.CD012854.pub2. PMID 36094829